CLINICAL TRIAL: NCT04329936
Title: Epidemiological Study on Mental Health of Migrant Population in the Retention Center of Geispolsheim
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7657
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Mental Health of Migrant Population
Keywords: Mental health; Psychiatric diseases; Migration; Retention center
MeSH Terms: conditions — Psychological Well-Being; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Retention center Geispolsheim population — All recently held individuals in the retention center can be included in the study after signing the information and consent protocol.

SUMMARY:
In 2019, the lack of studies about mental health of the detained population at retention centers in France is pointed out by the report of Controller-General for Places of Deprivation of Liberty. The aim of this study is to contribute to this relatively untouched field by describing which psychiatric pathologies are encountered in this population who went through migration and retention. Having a clearer picture of the situation can help to provide a more adapted psychiatric care in retention centers.

The results are expected to show a higher rate of psychiatric disease than in the general population including addiction to substance, anxiety disorder and post-traumatic stress disorder (PTSD).

ELIGIBILITY:
Inclusion Criteria:

* Any male person in the first week of detention at CRA Geispolsheim who gave their non-opposition to participation in the study.
* Information and consent protocol signed

Exclusion Criteria:

* Refuse to participate to the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The migrant population in the retention center of Geispolsheim is male migrants residing in France without authorization. Their retention is decided by the prefecture of Bas-Rhin and Haut-Rhin. The retention happens after custody or at the end of a term of imprisonment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Mini International Neuropsychiatric Interview validated and translated in the language used by the interviewed person. | 1 hour
  The interview is led by the investigator in the presence of a translator if necessary.

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided